CLINICAL TRIAL: NCT04617288
Title: Efficacy of SNAGs in the Management of Mechanical Neck Pain
Brief Title: SNAGs in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raj Nursing and Paramedical College (Other)
Responsible Party: Principal Investigator, Sharick Shamsi, Principal Investigator, Raj Nursing and Paramedical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RajNursingParamedicalC
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Ultrasonic Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to group A receiving conventional Physiotherapy plus SNAGs and group B receiving conventional Physiotherapy plus ultrasound.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mean and standard deviations of age and height between group A and B (Experimental): 100 subjects with a mean age of 30.82±6.75 (group A, 31.42±6.67; group B, 30.82±6.82) ranging from 20 to 45 years, with a mean height of 165.52±7.85 (group A, 164.92±7.79; group B, 166.12±7.87) centimeters
  Interventions: Other: Ultrasound Therapy, SNAGs
- Between group comparison of VAS, NDI and ROM (Experimental): VAS, NDI and Neck ROM between two groups were compared at pretest (0 day) and posttest (end of two weeks)
  Interventions: Other: Ultrasound Therapy, SNAGs

INTERVENTIONS:
Other: Ultrasound Therapy, SNAGs
  Other Names: Hot Pack, Exercise

SUMMARY:
Neck pain is second largest cause of disability worldwide. Chronic neck pain prevalence is 14% which is somewhat higher in females as compared to males. In India reported prevalence is 6%. Therapeutically, neck pain is managed by physiotherapists using rest, stretching and strengthening exercises, educating patient, and intense proprioception and positional exercises.

DETAILED DESCRIPTION:
To determine the evidences for the efficacy of SNAGs in the Management of Mechanical Neck Pain.

100 patients [Age group 25-45 yrs] who were diagnosed with neck pain, with onset ˃1-3 months (chronic) were randomly assigned to group A receiving conventional Physiotherapy plus SNAGs and group B receiving conventional Physiotherapy plus ultrasound.

Subjects in-group A that received conventional Physiotherapy plus SNAGs showed greater Improvement in pain and range of motion compared with the conventional Physiotherapy plus ultrasound group on 2nd week compared with pretreatment.

The result of study suggests that both SNAGs and Ultrasound groups improves the symptoms of neck pain. Ultrasound group improved the pain symptoms but was too small to reach satisfactory outcome for patients. Based on these results conventional Physiotherapy plus SNAGs should be the treatment of choice for neck pain rather than conventional Physiotherapy plus Ultrasound .

ELIGIBILITY:
Inclusion criteria

* Age group between 20- 45 years.
* Both Gender male and female.
* Individuals having localized pain or stiffness in spine or both combined b/w C3 to C7 without upper limbs radiculopathy.
* Pain reported on VAS score ˃3 in neck region.
* Patients agree to sign written consent form.

Exclusion Criteria Patients were excluded if they were diagnosed with following conditions for ˃6 months:

* T.B, carcinoma, heart disease, osteoporosis.
* Neural disorders due to PIVD.
* Any trauma or localized infection in neck region.
* Upper MND, cervical stenosis, metabolic diseases in bone and joint.
* Hyper flexibility
* Open sores,
* Ongoing radiotherapy, chemotherapy, steroid therapy or anticoagulants.
* Psychiatric diseases such as phobia/obsession, depression.
* Allergy to hot pack
* Patients with history of surgery in cervical spine region with in a year.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2015-08-25 (Actual); Study Completion 2015-08-25 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 2 weeks
  Visual analog scale is a subjective outcome measurement where patients judge the intensity of their pain on a scale of 0-10, which is in the form of a 10cm straight line. On this 0-10 scale, zero denotes no pain and ten denotes severe pain intensity.
Neck Range of motion | 2 weeks
  Range of motion of the cervical spine measured by bubble inclinometer. It consists of a 360-degree scale with a fluid filled circular tube containing a small air bubble. It is a gravity dependent Goniometer, which uses the gravity's effect on fluid level to measure joint position and motion.

SECONDARY OUTCOMES:
Neck disability Index | 2 weeks
  Neck disability Index contains 10 items, seven related to activities of daily living, two related to pain, and one item related to concentration. Each item is scored ranging from 0 (no pain or disability) to 5 (severe pain and disability); and the total score is expressed as a percentage, with higher scores corresponding to greater disability.

IPD SHARING:
Plan to Share IPD: No